CLINICAL TRIAL: NCT02583243
Title: Project BEST: Buprenorphine Entry Into Substance Abuse Treatment
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0504027630_B; SAMHSA TCE/HIV 15767
Record Dates: First submitted 2008-06-05; First posted 2015-10-22 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Opioid-related Disorders; HIV Infections; Hepatitis C, Chronic; Depression
Keywords: Opioid dependence; HIV/AIDS; Hepatitis C; Severe mental illness; Injection Drug Use
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections; Hepatitis C, Chronic; Depression; Acquired Immunodeficiency Syndrome; Hepatitis C; Mental Disorders | interventions — Buprenorphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: MET/CBT based individualized counseling — Manualized counseling with the first four week being MET followed by 8 weeks of CBT
Drug: Buprenorphine — Target dose in stabilization is 16 mg of buprenorphine to be taken sublingually once daily.

SUMMARY:
Project BEST is a clinical project funded by the Substance Abuse and Mental Health Services Administration (SAMHSA) to increase treatment to opiate dependent patients with mental illness in New Haven, CT and to prospectively follow everyone enrolled in buprenorphine care for as long as the individual takes buprenorphine to track the success of buprenorphine for the maintenance of opiate dependence.

DETAILED DESCRIPTION:
The investigators propose to create a prospective cohort that will track outcomes for an opiate dependent population on buprenorphine maintenance. Individuals who have already decided to undergo buprenorphine treatment in Project BEST will be invited to participate in the following data collection process. The investigators propose the following series of data collection to assess clients during their time in the cohort:

GPRA, supplemental instrument, ASI, SCID, COWS, Urine toxicology.

Patients who are enrolled will enter a standardized, manual based weekly counseling regimen. Urine toxicology will be performed a minimum of twice monthly, but will not occur at the same times monthly to decrease the probability of sampling error.

This is a prospective cohort to follow a group of individuals on buprenorphine treatment. The goal of this prospective cohort is to generate thoughtful observations. Specific items of interest which will be compared with age, race matched historical controls on methadone will be:

1. Changes in addiction severity over treatment time
2. Changes in sexual risk behaviors and injection practices
3. Improvements in urine toxicology
4. Co-occurring mental illness

ELIGIBILITY:
Inclusion Criteria:

* Opiate dependent by DSM IV criteria - to be determined by clinician - on buprenorphine through the Project BEST Program.

Exclusion Criteria:

* Inability to adhere to study instruments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort of opioid dependent patients at risk for HIV or with HIV seeking treatment with buprenorphine. Subjects may have severe mental illness and other co-morbid medical conditions.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University AIDS Program
Locations (1):
- Yale University, New Haven, Connecticut, United States